CLINICAL TRIAL: NCT06108297
Title: Effect of Low-dose Lithium Therapy on Long COVID Symptoms: an Open-label, Dose-finding Study.
Brief Title: Lithium Long COVID Dose-finding Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Thomas Guttuso, Professor of Neurology, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007796
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lithium (Experimental): Lithium capsules titrated to 30-45mg/day based on individual patient subjective benefits and tolerability.
  Interventions: Dietary Supplement: Lithium

INTERVENTIONS:
Dietary Supplement: Lithium — Elemental lithium as lithium aspartate.

SUMMARY:
This open-label study will assess if lithium dosages of 30-45mg/day are associated with greater symptomatic benefit than dosages of 10-15mg/day previously assessed among 50 patients with long COVID.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled from November 2022-July 2023 in lithium long COVID clinical trial at UB.
2. Reports bothersome fatigue and/or brain fog while not taking lithium or, reports satisfactory benefit to these symptoms while taking lithium.
3. Fatigue Severity Scale (FSS) score ≥28 or Brain Fog Severity Scale (BFSS) score ≥28 at baseline or; FSS <28, BFSS <28 and PGIC at Visit 1 of "much improved" or "very much improved" while taking lithium.
4. Did not "respond" to placebo therapy, based on the responder analyses outlined in the Preliminary data section above, defined as a ≥18-point reduction FSS or ≥15-point reduction in BFSS from baseline to the end-of-double-blind study phase while receiving placebo therapy.

Exclusion Criteria:

1. Fever or signs of acute infection in last 4 weeks.
2. COVID vaccine administered within 4 weeks. No change in any psychoactive or steroid medications for ≥30 days.
3. Plan to change a psychoactive, steroid or diuretic medication in next 5 weeks.
4. History of heart attack or stroke within the previous year.
5. Active medical, psychiatric or social problem that would interfere with completing the study procedures in the opinion of the investigator.
6. Daily NSAID use.
7. Pregnant or nursing or planning to get pregnant over the next 11 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale (FSS) | Baseline to end-of-titration (up to 11 weeks)
  7-item scale. Score range 1-49 with higher values signifying worse outcome
Brain Fog Severity Scale (BFSS) | Baseline to end-of-titration (up to 11 weeks)
  7-item scale. Score range 1-49 with higher values signifying worse outcome

SECONDARY OUTCOMES:
Well Being Scale | Baseline to end-of-titration (up to 11 weeks)
  Single-item question. Score range 0-10 with higher values signifying better outcome.
Short Form-12 Health Survey | Baseline to end-of-titration (up to 11 weeks)
  12-item quality of life scale. Score range 0-100 for both the Physical Component Score and the Mental Component Score with higher values signifying better outcomes.
FSS scores in those with FSS score ≥28 at baseline | Baseline to end-of-titration (up to 11 weeks)
  7-item scale. Score range 1-49 with higher values signifying worse outcome
BFSS scores in those with FSS score ≥28 at baseline | Baseline to end-of-titration (up to 11 weeks)
  7-item scale. Score range 1-49 with higher values signifying worse outcome
Modified Fatigue Impact Scale | Baseline to end-of-titration (up to 11 weeks)
  21-item scale. Score range 0-84 with higher values signifying worse outcome
Perceived Deficits Questionnaire, 5-Item Version | Baseline to end-of-titration (up to 11 weeks)
  5-item scale. Score range 1-20 with higher values signifying worse outcome
Beck Depression Inventory-II | Baseline to end-of-titration (up to 11 weeks)
  21-item scale. Score range 0-63 with higher values signifying worse outcome
Generalized Anxiety Disorder Scale-2 | Baseline to end-of-titration (up to 11 weeks)
  2-item scale. Score range 0-6 with higher values signifying worse outcome
Headache and Body Pain Bother Scale | Baseline to end-of-titration (up to 11 weeks)
  2-item scale. Score range 2-10 with higher values signifying worse outcome
Insomnia Severity Index | Baseline to end-of-titration (up to 11 weeks)
  7-item scale. Score range 0-28 with higher values signifying worse outcome
Patient Global Impression of Change | End-of-titration (up to 11 weeks)
  Single-item scale. Score range 1-7 with higher values signifying better outcome
Desire to Continue Therapy Scale | End-of-titration (up to 11 weeks)
  Single-item scale. Score range 1-2 with higher value signifying better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- UBMD Neurology, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guttuso T Jr, Zhu J, Wilding GE. Lithium Aspartate for Long COVID Fatigue and Cognitive Dysfunction: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2436874. doi: 10.1001/jamanetworkopen.2024.36874. PMID 39356507